CLINICAL TRIAL: NCT02895867
Title: Effect of Consumption of Dairy Products on Glycemic Control, Body Weight and Cardiovascular Risk Factors in Patients With Type 2 Diabetes: A Randomized Controlled Clinical Study
Brief Title: Effect of Dairy Consumption on Glycemic Control, Body Weight and Cardiovascular Risk in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-04
Record Dates: First submitted 2016-05-04; First posted 2016-09-12 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Full fat dairy group (Experimental): Participants will receive nutritional counseling aiming to maintain body weight from a registered dietitian and will be instructed to include at least ≥3 servings of full fat dairy products into their diet
  Interventions: Other: Full fat dairy
- Low fat dairy group (Experimental): Participants will receive nutritional counseling aiming to maintain body weight from a registered dietitian and will be instructed to include at least ≥3 servings of low fat dairy products into their diet
  Interventions: Other: Low fat dairy
- Control group (Other): Participants will receive nutritional counseling aiming to maintain body weight from a registered dietician and will not be asked to include a specified amount or type of dairy products
  Interventions: Other: Control

INTERVENTIONS:
Other: Full fat dairy — Participants will receive nutritional counseling aiming to maintain body weight from a registered dietician and will be instructed to include at least ≥3 servings of full fat dairy products into their diet
  Arms: Full fat dairy group
Other: Low fat dairy — Participants will receive nutritional counseling aiming to maintain body weight from a registered dietician and will be instructed to include at least ≥3 servings of low fat dairy products into their diet
  Arms: Low fat dairy group
Other: Control — Participants will receive nutritional counseling aiming to maintain body weight from a registered dietician and will not be asked to include a specified amount or type of dairy products
  Arms: Control group

SUMMARY:
This is a randomized prospective clinical study in patients with type 2 diabetes to evaluate the effect of dairy products with full or low fat on glycemic control and cardio-metabolic risk factors in comparison to a regular diet.

DETAILED DESCRIPTION:
This is a randomized, controlled clinical study in which 108 subjects with type 2 diabetes will be randomized into 3 different groups:

Full fat dairy group (Group A): will receive nutritional counseling aiming to maintain body weight from a registered dietician and will be instructed to include at least ≥3 servings of full fat dairy products into their diet

Low fat dairy group (Group B): will receive nutritional counseling aiming to maintain body weight from a registered dietician and will be instructed to include at least ≥3 servings of low fat dairy products into their diet

Control group (Group C): will receive nutritional counseling aiming to maintain body weight from a registered dietician and will not be asked to include a specified amount or type of dairy products

Subjects in Groups A and B will be educated about different dairy products' serving sizes and fat content. Subjects in all 3 groups will be asked to record their daily intake of dairy products in a dedicated log book. Subjects randomized to groups A and B will be asked to only use only dairy products with either the full fat or and low (≤1%) fat dairy (≤1% fat content) content respectively. Purchase of the dairy products will be the responsibility of study subjects for which a subsidy of $500 (about $20/week for 24 weeks) will be provided for each subject. All study participants will also be asked to record their food intake for 3 days before each study visit in a 3-day food log.

ELIGIBILITY:
Inclusion Criteria:

* Having type 2 diabetes for at least three months prior to screening and treated with any antihyperglycemic medication
* A1C ≥7 %
* Consuming <3 servings of dairy products per day
* On stable dose of diabetes, blood pressure or cholesterol medications for 3 months
* Body weight is within 10% of current weight over the last 6 months before starting the study

Exclusion Criteria:

* Pregnancy or lactation
* Lactose intolerance
* Allergy to milk or any of its components
* Use of orlistat
* History of pancreatitis
* History of gastric bypass surgery or sleeve gastrectomy
* Active malignancy
* History of recent cardiovascular event
* Having a heart pacemaker
* Enrollment in other studies that may affect study outcomes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-05; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1C (A1C) | Baseline, 12 weeks and 24 weeks

SECONDARY OUTCOMES:
Change in body weight | Baseline, 12 weeks and 24 weeks
Change in total cholesterol | Baseline, 12 weeks and 24 weeks
Change in high-density lipoprotein (HDL) | Baseline, 12 weeks and 24 weeks
Change in low-density lipoprotein (LDL) | Baseline, 12 weeks and 24 weeks
Change in triglycerides | Baseline, 12 weeks and 24 weeks
Change in fasting plasma glucose | Baseline, 12 weeks and 24 weeks
Change in Homeostatic model assessment (HOMA) insulin resistance (IR) index after 24 weeks compared to baseline | Baseline, 12 weeks and 24 weeks
Change in body fat percentage | Baseline, 12 weeks and 24 weeks
Change in fat free mass | Baseline, 12 weeks and 24 weeks
Height in meters | Baseline
  Used in calculation of Body Mass Index
Change in total body water | Baseline, 12 weeks and 24 weeks
Change in waist circumference | Baseline, 12 weeks and 24 weeks
Change in trunk fat percentage | Baseline, 12 weeks and 24 weeks
Change in visceral fat level | Baseline, 12 weeks and 24 weeks
Change in blood pressure | Baseline, 12 weeks and 24 weeks
Change in c-reactive protein level | Baseline, 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Osama Hamdy, M.D., Ph.D., Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitri J, Tomah S, Mottalib A, Salsberg V, Ashrafzadeh S, Pober DM, Eldib AH, Tasabehji MW, Hamdy O. Effect of dairy consumption and its fat content on glycemic control and cardiovascular disease risk factors in patients with type 2 diabetes: a randomized controlled study. Am J Clin Nutr. 2020 Aug 1;112(2):293-302. doi: 10.1093/ajcn/nqaa138. PMID 32520346